CLINICAL TRIAL: NCT06705764
Title: Tezepelumab in the Treatment of Emergency Room Asthma in Adults (TERAA): A Phase 4 Double-Blinded, Parallel-Group, Randomized Control Trial With an Open Label Extension
Brief Title: Tezepelumab in the Treatment of Emergency Room Asthma in Adults (TERAA)
Acronym: TERAA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESR-22-22102
Record Dates: First submitted 2024-10-18; First posted 2024-11-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Severe Asthma
Keywords: Asthma; Severe Asthma; Asthma Exacerbation; Tezepelumab; Emergency deparment visits for asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Tezepelumab (Active Comparator): Tezepelumab 210 mg S/Q Q4W
  Interventions: Drug: Tezepelumab
- Placebo (Placebo Comparator): Matching Placebo S/Q Q4W
  Interventions: Drug: Placebo
- Tezepelumab Open Label (Other): Open-label extension study from Day 90 to Day 180 with Tezepelumab dosing at Day 90
  Interventions: Drug: Tezepelumab

INTERVENTIONS:
Drug: Tezepelumab — Tezepelumab 210 mg (1.91 ml) subcutaneous every 4 weeks. Randomized Control Trial 90 days with Tezepelumab/ Matching Placebo dosing on Day 0, Day 30 and Day 60.
  Open-label extension study from Day 90 to Day 180 with Tezepelumab dosing at Day 90
  Arms: Tezepelumab; Tezepelumab Open Label
Drug: Placebo — Placebo 1.91 ml subcutaneous every 4 weeks. Randomized Control Trial 90 days with Tezepelumab/ Matching Placebo dosing on Day 0, Day 30 and Day 60.
  Arms: Placebo

SUMMARY:
Adults with severe asthma may have sudden worsening shortness of breath that results in their going to Emergency Department for urgent care. Emergency Room visits for asthma management across Alberta have been reviewed and it has been found that adults frequently need to return for repeated worsening. This is a large drain on health care resources as well as being very distressing for individuals with asthma. Occasionally this results in admission to hospital and rarely may lead to death. People are often treated with steroids to try to prevent the need for Emergency Room visits even though steroid medications have many long term bad side effects.

A new medication for patients considered to have severe asthma has been recently approved by Health Canada. This medication, Tezepelumab, is a monthly injection and it helps control asthma in adults regardless of the underlying cause. The study will examine if starting Tezepelumab, compared with a placebo, in the Emergency Room will help settle symptoms of asthma and prevent future worsening requiring repeated Emergency Room visits or the need for courses of outpatient steroid medications.

DETAILED DESCRIPTION:
All patients with a physician-diagnosed history of asthma and a history of a moderate or severe exacerbation of asthma presenting to the Emergency Department (ED) with an acute exacerbation of asthma will be reviewed by a study coordinator. From this population, subjects with at least 3-month history of prescription for a high dose inhaled corticosteroid (ICS) plus a reliever medication such as a long-acting beta2 agonist (LABA), long-acting muscarinic antagonist (LAMA) or a leukotriene receptor antagonist (LRTA) will be approached for study enrolment while still within the ED. Following informed consent, subject will be randomized in a 1:1 ratio to either Tezepelumab 210 mg S/Q Q4W or to a marching placebo. The proportion of subjects returning to ED for an exacerbation of asthma by Day-90 will serve as the primary study outcome. After Day-90 subjects will be entered into an open-label study with all receiving Tezepelumab 210 mg S/Q Q4W. A key secondary outcome will be the proportion of subjects returning to ED for an exacerbation of asthma by Day-180. Other secondary outcomes will include Alarmin expression, ACQ-5, FEV1 as well as study drug safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female and/or male aged 18 to 55 years
3. History of physician-diagnosed asthma
4. All subjects will have been prescribed high dose inhaled corticosteroid (> 500 ug fluticasone propionate dry powder formulation equivalents total daily dose. See Appendix C) plus at least one second controller (LABA, LAMA or LTRA) for at least 3 months prior to enrolment.
5. Documented history of at least one moderate or severe asthma exacerbation in the past 12 months
6. Negative pregnancy test (urine or serum) for female subjects of childbearing potential.
7. Female subjects must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of study drug/matching placebo to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.
8. Subjects who are blood donors should not donate blood during the study and for 3 months following their last dose of study drug.
9. Subject willing and able to comply with study procedures

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
2. Previous enrolment in the present study
3. Participation in another clinical study with an investigational product during the last 6 months
4. Patients with a known hypersensitivity to Tezepelumab or any of the excipients of the product.
5. Patients who are admitted to hospital at screening.
6. Positive hepatitis C antibody hepatitis B virus surface antigen or hepatitis B virus core antibody, at screening.
7. Known to have tested positive for human immunodeficiency virus
8. Current smokers with a smoking history of > 10 pack-years. Current smokers with a smoking history of < 10 pack-years are permitted . Ex-smokers should not have a smoking history > 10 pack-years at screening. Participants who use e-cigarettes will also be excluded from the study.
9. Known history of drug or alcohol abuse within 1 year of screening
10. Any concomitant medications that are known to be associated with Torsades de Pointes or potent inducers of cytochrome P450 3A4 (CYP3A4).
11. History of QT prolongation associated with other medications that required discontinuation of that medication.
12. Congenital long QT syndrome.
13. Creatinine clearance <50 ml/min (calculated by Cockcroft-Gault formula, reference Appendix G).
14. For women only - currently pregnant (confirmed with positive pregnancy test) or breast feeding.
15. History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Subjects with atrial fibrillation controlled by medication are permitted.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who have moderate and severe exacerbations of asthma | 90 Days post-treatment
  Numbers of moderate and severe exacerbations at Day 90 post-treatment in subjects treated with standard care and S/Q Tezepelumab or treated with standard care and placebo

SECONDARY OUTCOMES:
Numbers of subjects returning to ED | 90 Days post-treatment
  Numbers of subjects returning to ED by Day-90 in those treated with standard care and S/Q Tezepelumab or treated with standard care and placebo.
Proportion of subjects returning to ED | 60 Days post-treatment
  Proportion of subjects returning to ED by Day-30 and Day-60 in those treated with standard care and S/Q Tezepelumab or treated with standard care and placebo.
Asthma control Questionnaire (ACQ-5) | 90 Days post-treatment
  ACQ-5 at Day-90 in subjects treated with standard care and S/Q Tezepelumab or treated with standard care and placebo ACQ-5 greater than 1.5 units in subjects treated with standard care and S/Q Tezepelumab or treated with standard care and placebo ACQ-5 less than 0.75 units in subjects treated with standard care and S/Q Tezepelumab or treated with standard care and placebo
  ACQ (Asthma Control Questionnaire). Each question is scored on a scale of 0 to 6, with 0 representing excellent control and 6 representing extremely poor control. The final score is the mean of the five responses.
TSLP levels | Day 1
  TSLP levels at the time of ED presentation
IL-25 levels | Day 1
  IL-25 levels at the time of ED presentation
Il-33 levels | Day 1
  IL-33 levels at the time of ED presentation

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by an intensity rating scale | Through study completion, an average of 180 days
  To evaluate the safety and tolerability of Tezepelumab in relation to Placebo the results from laboratory tests and vital signs will be assessed to determine treatment-related adverse events.
Nasal brushing expressions of TSLP(Exploratory Outcome) | Day-30, 90 and 180 post ED visit
  Nasal brushing expressions of TSLP
Measure ACQ-5 at selected time-points (Exploratory Outcome) | Day-30, 90 and 180 post ED visit
  Compare time course of ACQ-5 following discharge from ED in subjects treated with standard care and S/Q Tezepelumab or treated with standard care and placebo at Day-30, 90 and 180 post ED visit.
  1. Compare frequency of uncontrolled subjects (ACQ-5 greater than 1.5 units) in subjects treated with standard care and S/Q Tezepelumab or treated with standard care and placebo at Day-30 and 180.
  2. Compare frequency of well-controlled subjects (ACQ-5 less than 0.75 units) in subjects treated with standard care and S/Q Tezepelumab or treated with standard care and placebo at Day-30 and 180.
  ACQ (Asthma Control Questionnaire). Each question is scored on a scale of 0 to 6, with 0 representing excellent control and 6 representing extremely poor control. The final score is the mean of the five responses.
Measure pre-bronchodilator FEV1 at selected time points (exploratory outcome) | Day 30, 90 and 180 days post ED visit
  Compare time course of lung function, assessed as in-laboratory FEV1, following discharge from ED in subjects treated with standard care and S/Q Tezepelumab or treated with standard care and placebo at 30, 90 and 180 days post ED visit.
Measure TSLP expression at various time points Peripheral blood eosinophil counts FeNO Serum IgE (Exploratory Outcome) | Day 1
  Correlate acute asthma severity with TSLP expression during ED visit
  1. Compare TSLP expression during ED visit in subjects with Type 2 asthma and non-Type 2 asthma
  2. Measure cell and plasma expression of TSLP, IL-25 and IL-33 in subjects presenting to ED following an acute asthma exacerbation obtained from nasopharyngeal and plasma samples.
FeNO will be tested at selected time-points (Exploratory Outcome) | Day 30, 90 and 180 post ED visit
  Compare time course of FeNO following discharge from ED in subjects treated with standard care and S/Q Tezepelumab or treated with standard care and placebo at Day-30, 90 and 180 post ED visit.
Nasal brushing expressions of IL-33 (Exploratory Outcome) | Day-30, 90 and 180 post ED visit
  Nasal brushing expressions of IL-33
Nasal brushing expressions of IL-25 (Exploratory Outcome) | Day-30, 90 and 180 post ED visit
  Nasal brushing expressions of IL-25
Measure pre-bronchodilator PEF at selected time points (exploratory outcome) | Day-30, 90 and 180 post ED visit
  Compare time course of lung function, assessed as at home PEF, following discharge from ED in subjects treated with standard care and S/Q Tezepelumab or treated with standard care and placebo at 30, 90 and 180 days post ED visit.

CONTACTS AND LOCATIONS:
Overall Officials: Irvin Mayers, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Sturgeon Community Hospital, St. Albert, Alberta
  - University of Alberta, Edmonton, Ca-ab

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhao W, Weng Y. Block urn design - a new randomization algorithm for sequential trials with two or more treatments and balanced or unbalanced allocation. Contemp Clin Trials. 2011 Nov;32(6):953-61. doi: 10.1016/j.cct.2011.08.004. Epub 2011 Aug 22. PMID 21893215
- [Result] Wang W, Li Y, Lv Z, Chen Y, Li Y, Huang K, Corrigan CJ, Ying S. Bronchial Allergen Challenge of Patients with Atopic Asthma Triggers an Alarmin (IL-33, TSLP, and IL-25) Response in the Airways Epithelium and Submucosa. J Immunol. 2018 Oct 15;201(8):2221-2231. doi: 10.4049/jimmunol.1800709. Epub 2018 Sep 5. PMID 30185520
- [Result] Osborne NJ, Alcock I, Wheeler BW, Hajat S, Sarran C, Clewlow Y, McInnes RN, Hemming D, White M, Vardoulakis S, Fleming LE. Pollen exposure and hospitalization due to asthma exacerbations: daily time series in a European city. Int J Biometeorol. 2017 Oct;61(10):1837-1848. doi: 10.1007/s00484-017-1369-2. Epub 2017 May 12. PMID 28500390
- [Result] Mayers I, Randhawa A, Qian C, Talukdar M, Soliman M, Jayasingh P, Johnston K, Bhutani M. Asthma-related emergency admissions and associated healthcare resource use in Alberta, Canada. BMJ Open Respir Res. 2023 Oct;10(1):e001934. doi: 10.1136/bmjresp-2023-001934. PMID 37914234
- [Result] Khatri SB, Iaccarino JM, Barochia A, Soghier I, Akuthota P, Brady A, Covar RA, Debley JS, Diamant Z, Fitzpatrick AM, Kaminsky DA, Kenyon NJ, Khurana S, Lipworth BJ, McCarthy K, Peters M, Que LG, Ross KR, Schneider-Futschik EK, Sorkness CA, Hallstrand TS; American Thoracic Society Assembly on Allergy, Immunology, and Inflammation. Use of Fractional Exhaled Nitric Oxide to Guide the Treatment of Asthma: An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2021 Nov 15;204(10):e97-e109. doi: 10.1164/rccm.202109-2093ST. PMID 34779751
- [Result] Juniper EF, Bousquet J, Abetz L, Bateman ED; GOAL Committee. Identifying 'well-controlled' and 'not well-controlled' asthma using the Asthma Control Questionnaire. Respir Med. 2006 Apr;100(4):616-21. doi: 10.1016/j.rmed.2005.08.012. Epub 2005 Oct 13. PMID 16226443
- [Result] Juniper EF, Svensson K, Mork AC, Stahl E. Measurement properties and interpretation of three shortened versions of the asthma control questionnaire. Respir Med. 2005 May;99(5):553-8. doi: 10.1016/j.rmed.2004.10.008. Epub 2004 Nov 26. PMID 15823451
- [Result] Hsu SC, Chang JH, Lee CL, Huang WC, Hsu YP, Liu CT, Jean SS, Huang SK, Hsu CW. Differential time-lag effects of ambient PM2.5 and PM2.5-bound PAHs on asthma emergency department visits. Environ Sci Pollut Res Int. 2020 Dec;27(34):43117-43124. doi: 10.1007/s11356-020-10243-y. Epub 2020 Jul 29. PMID 32729038
- [Result] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Result] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Result] Berger VW, Bejleri K, Agnor R. Comparing MTI randomization procedures to blocked randomization. Stat Med. 2016 Feb 28;35(5):685-94. doi: 10.1002/sim.6637. Epub 2015 Sep 3. PMID 26337607
- [Result] Baren JM, Boudreaux ED, Brenner BE, Cydulka RK, Rowe BH, Clark S, Camargo CA Jr. Randomized controlled trial of emergency department interventions to improve primary care follow-up for patients with acute asthma. Chest. 2006 Feb;129(2):257-265. doi: 10.1378/chest.129.2.257. PMID 16478839
- See also: Global Strategy for Asthma Management and Prevention, Global Initiative for Asthma (GINA). Updated 2024 — http://www.ginasthma.org/